CLINICAL TRIAL: NCT06205134
Title: A Study to Compare the Bioavailability of Epinephrine Following a Single Nasal Dose of FMXIN002 Microspheres Powder 3.6mg, and 4mg With EpiPen 0.3mg Intramuscular Injection in Healthy Adults
Brief Title: Comparative Bioavailability of Intranasal Epinephrine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nasus Pharma (Industry)
Collaborators: Hadassah Medical Organization (Other); Medistat Ltd., Israel (Industry); Pharma Medica Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP-006-Epinephrine
Record Dates: First submitted 2023-12-18; First posted 2024-01-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-03

CONDITIONS: Anaphylaxis; Anaphylactic Reaction
Keywords: Anaphylaxis; Epinephrine; Nasal; spray; Pharmacokinetics
MeSH Terms: conditions — Anaphylaxis | interventions — Epinephrine

STUDY DESIGN:
Intervention Model Description: To evaluate the comparative bioavailability and pharmacodynamic response between:
  A. Epinephrine injection, USP auto-injector 0.3 mg for intramuscular (IM) injection B. FMXIN002 epinephrine microspheres powder for nasal application, 3.6 mg and C. FMXIN002 epinephrine microspheres powder for nasal application, 4 mg and after a single-dose administration to healthy adults
  Secondary Objective:
  To evaluate the safety and tolerability of the study treatments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 6 Healthy volunteers, sequence ABC (Experimental): Three drug administrations to each subject, each administration on a separate day.
  treatment order: A B C
  Interventions: Drug: A: Epinephrine injection; Drug: B: FMXIN002 3.6mg; Drug: C: FMXIN002 4.0mg
- 6 Healthy volunteers, sequence BAC (Experimental): Three drug administrations to each subject, each administration on a separate day.
  treatment order: B A C
  Interventions: Drug: A: Epinephrine injection; Drug: B: FMXIN002 3.6mg; Drug: C: FMXIN002 4.0mg

INTERVENTIONS:
Drug: A: Epinephrine injection — Autoinjector for intramuscular, single-use, 0.3mg
  Other Names: EpiPen
Drug: B: FMXIN002 3.6mg — Nasus Pharma nasal powder spray 3.6 mg, single use in one nostril
  Other Names: Epinephrine Nasal Product
Drug: C: FMXIN002 4.0mg — Nasus Pharma nasal powder spray 4.0 mg, single use in one nostril
  Other Names: Epinephrine Nasal Product

SUMMARY:
A Study to Compare the Bioavailability of Epinephrine following a Single Nasal Dose of FMXIN002 Microspheres Powder 3.6 mg, and 4mg with EpiPen 0.3mg Intramuscular Injection in Healthy Adults

DETAILED DESCRIPTION:
An open-label trial in 12 healthy adults. FMXIN002 (3.6 mg and 4.0 mg) will be administered intranasally to healthy adults and compared to IM (0.3mg, EpiPen) by Epinephrine pharmacokinetics, pharmacodynamic response and clinical safety.

(https://my.health.gov.il/CliniTrials/Pages/MOH_2023-07-01_012776.aspx.)

ELIGIBILITY:
Inclusion Criteria:

* 1) Non-smoking, male and female subjects from 18 to 55 years of age. 2) BMI ≥18 < 30 kg/m2. 3) Females may be of childbearing or non-childbearing potential:

  * Childbearing potential:

    o Physically capable of becoming pregnant, must be willing to use acceptable effective methods of contraception
  * Non-childbearing potential:

    * Surgically sterile
    * Postmenopausal (no menstrual period for at least 12 consecutive months without any other medical cause).

      4) Able to tolerate venipuncture. 5) Be informed of the nature of the study and give written consent prior to any study procedure.

      6) Willing and being able to remain in the clinic for the entire duration of the confinement period.

      7) Have good intravenous access on both arms and hands.

Exclusion Criteria:

* 1) Known history or presence of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, ischemic heart disease or Arteriosclerosis or cardiovascular disease, autoimmune disease, or Raynaud Phenomenon and any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.

  1. Known history or presence of hypersensitivity or idiosyncratic reaction to epinephrine, sulfite, other excipients of epinephrine auto-injector, or any other drug substances with similar activity.
  2. Known history or presence of clinically significant lactose, galactose, or fructose allergy
  3. Known history or presence of any food allergy.
  4. Presence of nostril or septum piercing.
  5. Presence of abnormal nasal anatomy (e.g., polyps, unilateral or bilateral abnormalities of the nares, nasal turbinates, or septum including deviated septum).
  6. History of nasal surgery.
  7. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption other than oral contraceptives.
  8. History of drug or alcohol addiction requiring treatment or positive alcohol breath test at check-in.
  9. Any acute illness (e.g. cold, acute infection) which is considered significant by the Investigator and that has not resolved within 7 days before the first drug administration.
  10. Positive test result for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
  11. Positive test result for urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, phencyclidine, and tricyclic antidepressants) or urine cotinine.
  12. Inability to communicate well with the Investigators and staff
  13. Non-cooperative or unwilling to sign consent form or unwilling to attend scheduled clinic visits and/or comply with the study protocol.
  14. Use of tobacco or nicotine-containing products within 6 months prior to drug administration.
  15. Females who:

      * Have discontinued or changed the use of implanted, intrauterine, intravaginal, or injected hormonal contraceptives within 6 months prior to drug administration;
      * Have discontinued or changed the use of oral or patch hormonal contraceptives within 1 month prior to drug administration;
      * Are pregnant (Urine hCG consistent with pregnancy); or
      * Are lactating.
  16. Donation or loss of whole blood (including clinical trials):

      * ≥50 mL and <500 mL within 30 days prior to drug administration;
      * ≥500 mL within 56 days prior to drug administration.
  17. Participation in a clinical trial that involved administration of an investigational medicinal product within 30 days prior to drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results.
  18. On a special diet within 30 days prior to drug administration (e.g., liquid, protein, raw food diet).
  19. Have had a tattoo or body piercing within 30 days prior to drug administration.
  20. Have clinically significant findings in vital signs measurements at screening.
  21. Systolic blood pressure increase or decrease in value by more than 20 mmHg and/or diastolic blood pressure decrease in value by more than 10 mmHg, from supine or sitting to standing position during orthostatic blood pressure measurement taken at screening.
  22. Have clinically significant findings in a 12-lead ECG.
  23. Have clinically significant abnormal laboratory values and hemoglobin <135 g/L for males or <120 g/L for females at screening.
  24. Have significant diseases at screening.
  25. Have clinically significant findings from a physical examination.
  26. Use of the following drugs within 14 days prior to drug administration:

      * Alpha-adrenergic blocking drugs (e.g., phentolamine);
      * Anti-arrhythmics;
      * Beta-adrenergic blocking drugs (e.g., propranolol);
      * Cardiac glycosides;
      * Diuretics;
      * Drugs having effect on cytochrome P450 (CYP450);
      * Enzyme-altering drugs (e.g., barbiturates, phenothiazines, cimetidine, carbamazepine, etc.);
      * Enzyme-modifying drugs known to induce/inhibit hepatic drug metabolism;
      * Ergot alkaloids;
      * Levothyroxine sodium;
      * Monoamine oxidase inhibitors;
      * Oral or topical corticosteroids;
      * Phenylephrine;
      * Reserpine-type or clonidine-type antihypertensives;
      * Sodium cromoglycate; or
      * Tricyclic antidepressants.
  27. Use of the following drugs within 7 days prior to drug administration:

      * Nasal decongestants;
      * Nonsteroidal anti-inflammatory drugs (NSAIDs); or
      * Oral or topical antihistamines.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Bioavailability of Epinephrine | -1 to 2 hours post dose
  Plasma level of Epinephrine
Blood pressure | -1 to 4 hours post dose
  Pharmacodynamic response
Heart rate | -1 to 4 hours post dose
  Pharmacodynamic response
Respiratory rate | -1 to 4 hours post dose
  Pharmacodynamic response

SECONDARY OUTCOMES:
12-lead electrocardiogram | -2 up to 1 hour post dose
  Safety
Adverse events | through study completion, an average of 3 weeks
  Safety
Nasal Mucosa health status | -1 hour until end of each dosing day, an average 3 weeks.
  * Nasal cavity examination by physician, recorded on a severity scale
  * Nasal and Non-Nasal Questionnaire of symptomes, completed by the subjects, using a severity scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, Professor, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Clinical Pharmacology Unit, Hadassah Medical Center, Ein Karem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: First-in-class intranasal epinephrine spray for anaphylaxis: Dose finding clinical study — https://doi.org/10.1016/j.jacig.2025.100487